CLINICAL TRIAL: NCT05305989
Title: Extended Treatment and Follow-up of Subjects Treated With Belumosudil in Study KD025-208 or Study KD025-213
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LTS17660; KD025-217 (Other: Sanofi Identifier); U1111-1279-2612 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-02-02; First posted 2022-03-31 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: belumosudil 200 mg QD (Experimental): The assigned arm is per the previous study KD025-213 or study KD025-208
  Interventions: Drug: Belumosudil 200 mg QD
- Arm B: belumosudil 200 mg BID (Experimental): The assigned arm is per the previous study KD025-213 or study KD025-208
  Interventions: Drug: Belumosudil 200 mg BID
- Arm C: belumosudil 400 mg QD (Experimental): The assigned arm is per the previous study KD025-213 or study KD025-208
  Interventions: Drug: Belumosudil 400 mg QD

INTERVENTIONS:
Drug: Belumosudil 200 mg QD — Belumosudil is an orally available Rho-associated protein kinase-2 (ROCK2) selective inhibitor.
  Other Names: REZUROCK
  Arms: Arm A: belumosudil 200 mg QD
Drug: Belumosudil 200 mg BID — Belumosudil is an orally available Rho-associated protein kinase-2 (ROCK2) selective inhibitor.
  Other Names: REZUROCK
  Arms: Arm B: belumosudil 200 mg BID
Drug: Belumosudil 400 mg QD — Belumosudil is an orally available Rho-associated protein kinase-2 (ROCK2) selective inhibitor.
  Other Names: REZUROCK
  Arms: Arm C: belumosudil 400 mg QD

SUMMARY:
Extended Treatment and Follow-up of Subjects Treated with Belumosudil in Study KD025-208 or Study KD025-213

DETAILED DESCRIPTION:
This is a Phase 2, open-label, long-term treatment and follow-up study in subjects with cGVHD who have been previously treated with belumosudil in Study KD025-208 or Study KD025-213. Subjects will not be screened. Subjects who have signed the informed consent form will be enrolled in Study KD025-217 if they have met 1 of the following conditions:

* Actively receiving belumosudil or in long-term follow-up (LTFU) in Study KD025-208 or Study KD025-213
* Enrolled in the Companion Study as specified in Study KD025-213 Amendment 2 and received at least 6 months of treatment or is in LTFU

Approximately 20 Study Centers will participate with approximately 70 subjects participating overall.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have been treated with belumosudil for at least 1 of the following:

* Actively receiving belumosudil on Study KD025-208 or Study KD025-213
* Is in Long-term Follow-up (LTFU) on Study KD025-208 or Study KD025-213. Long-term Follow-up will be defined as the period after ending treatment with belumosudil and until a FFS event occurs.
* Adult enrolled in the Companion Study under KD025-213 Amendment 2 (01 June 2020) and has received at least 6 months of treatment of belumosudil or is in LTFU

Exclusion Criteria:

* Female subject who is pregnant or breastfeeding
* Subject considered unlikely to adhere to treatment and/or follow protocol in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope Site Number : 050, Duarte, California
  - Stanford Cancer Center Site Number : 108, Stanford, California
  - Washington University School of Medicine Site Number : 125, St Louis, Missouri
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center Site Number : 132, Pittsburgh, Pennsylvania
  - South Austin Medical Center Site Number : 091, Austin, Texas
  - MD Anderson Cancer Center Site Number : 057, Houston, Texas
  - Texas Transplant Institute Site Number : 079, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center Site Number : 052, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 8 sites in the United States from 23-Feb-2022 to 06-Jun-2024.
Pre-assignment Details: A total of 23 participants with chronic graft-versus-host-disease (cGVHD) who were previously treated with belumosudil in study KD025-208 (NCT02841995) or study KD025-213 (NCT03640481) were enrolled in this study.
Groups:
- Belumosudil 200 mg QD: Participants received belumosudil 200 milligrams (mg) tablet orally once a day (QD) until cGVHD progression, unacceptable toxicity or up to 2 years at the discretion of the Investigator.
- Belumosudil 200 mg BID: Participants received belumosudil 200 mg tablet orally twice a day (BID) until cGVHD progression, unacceptable toxicity or up to 2 years at the discretion of the Investigator.
- Belumosudil 400 mg QD: Participants received belumosudil 400 mg tablet orally QD until cGVHD progression, unacceptable toxicity or up to 2 years at the discretion of the Investigator.
Period: Overall Study
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Started | 13 | 9 | 1
Completed | 0 | 0 | 0
Not Completed | 13 | 9 | 1
Not completed — Other | 3 | 2 | 0
Not completed — Sponsor decision | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Investigator decision | 1 | 2 | 0
Not completed — Progression of cGVHD (progression requiring addition of new systemic therapy for cGVHD) | 3 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Enrolled but never dosed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants enrolled in the study.
Groups:
- Belumosudil 200 mg QD: Participants received belumosudil 200 mg tablet orally QD until cGVHD progression, unacceptable toxicity or up to 2 years at the discretion of the Investigator.
- Belumosudil 200 mg BID: Participants received belumosudil 200 mg tablet orally BID until cGVHD progression, unacceptable toxicity or up to 2 years at the discretion of the Investigator.
- Total: Total of all reporting groups
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD | Total
Number analyzed (Participants) | 13 | 9 | 1 | 23
Age, Customized [Count of Participants; unit: Participants]
  24-74 years | 13 | 9 | 1 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 9 | 7 | 0 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 12 | 9 | 1 | 22
  Not reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Response (DOR)
Description: DOR is defined as time from first documentation of response to time of first documentation of deterioration from best response (e.g., complete response [CR] to partial response [PR], or PR to Lack of response [LR]). As per the 2014 National Institutes of Health (NIH) Consensus Development Project for clinical trials in cGVHD criteria: CR was defined as resolution of all manifestations of cGVHD in each organ or site.PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site.LR included response status of mixed, unchanged, or progression.Mixed LR was defined as complete or partial response in at least 1 organ accompanied by progression in another organ. Unchanged LR was defined as outcomes that did not meet criteria for CR, PR, progression or mixed response. Progression LR was defined as progression in at least 1 organ or site without a response in any other organ or site. Confidence interval (CI) is calculated using Kaplan-Meier method.
Time Frame: At Baseline (Day 1), Month 3 and every 3 months thereafter (+/-14 days), up to 23 months
Population: Responder population included participants in the full analysis set that achieved a partial or complete response at any post-baseline response assessment. Only those participants who achieved CR or PR are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 8 | 8 | 0
months | NA [5.55 to NA] — NA indicates that median and upper limit of confidence interval (CI) were not estimable due to insufficient number of participants with events at study closure. | NA [5.78 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. |

2. Primary Outcome: Number of Participants With a >=7 Point Reduction (7PtR) From Baseline and >=7 Point Reduction From Baseline on 2 Consecutive Post-Baseline Assessments as Assessed by Lee Symptom Scale (LSS)
Description: The questionnaire asked participants to indicate the degree of bother that they experienced due to symptoms in 7 domains potentially affected by cGVHD. It consists of 30 items of 7 domains: skin, eyes and mouth, breathing, eating and digestion, muscles and joints, energy, and mental and emotional. Each question was rated/scored as 0-not at all, 1-slightly, 2-moderately, 3-quite a bit, 4-extremely with lower values representing better outcome. A domain score was calculated for each domain by taking the mean of all items completed if more than 50% were answered and normalizing to a 0 to 100 scale. A total score was calculated as average of all non-missing domain scores if more than 50% of them were non-missing, ranged from 0-100. A higher score indicated more bothersome symptoms. A 7-point difference on the total score of cGVHD symptom scale was found to be clinically meaningful.
Time Frame: Baseline (Day 1) up to 23 months
Population: The full analysis set included all participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
Participants
  >=7PtR From Baseline | 8 | 2 | 0
  >=7PtR From Baseline on 2 Consecutive Post-Baseline Assessment | 8 | 1 | 0

3. Primary Outcome: Duration of >=7 Point Reduction as Assessed by Lee Symptom Scale
Description: The questionnaire asked participants to indicate the degree of bother that they experienced due to symptoms in 7 domains potentially affected by cGVHD. It consisted of 30 items of 7 domains: skin, eyes and mouth, breathing, eating and digestion, muscles and joints, energy, and mental and emotional. Each question was rated/scored as 0-not at all, 1-slightly, 2-moderately, 3-quite a bit, 4-extremely with lower values representing better outcome. A domain score was calculated for each domain by taking the mean of all items completed if more than 50% were answered and normalizing to a 0 to 100 scale. A total score was calculated as average of all non-missing domain scores if more than 50% of them were non-missing, ranged from 0-100. A higher score indicated more bothersome symptoms. A 7-point difference on the total score of cGVHD symptom scale was found to be clinically meaningful. Mean of duration of >=7PtR is presented.
Time Frame: Baseline (Day 1) up to 23 months
Population: The full analysis set included all participants enrolled in the study. Only those participants with >=7PtR from Baseline are included in the analysis.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 8 | 2 | 0
weeks | 67.2 (26.8) | 49.5 (54.2) |

4. Primary Outcome: Time to Next Treatment (TTNT)
Description: The TTNT was measured as the time from first treatment to the time of new systemic cGVHD treatment, censored by last response assessment or long term follow up assessment, whichever was the latest and available. TTNT was analyzed by the Kaplan-Meier survival method.
Time Frame: At Baseline (Day 1), Month 3 and every 3 months thereafter (+/-14 days), up to 23 months
Population: The full analysis set included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
months | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. | NA [5.14 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure.

5. Primary Outcome: Failure-Free Survival (FFS)
Description: FFS was defined as the absence of new cGVHD systemic therapy, non-relapse mortality and recurrent malignancy (i.e. underlying disease) and was censored by last response assessment or long term follow up assessment, whichever was the latest and available. Kaplan-Meier method was used for the analysis.
Time Frame: At Baseline (Day 1), Month 3 and every 3 months thereafter (+/-14 days), up to 23 months
Population: The full analysis set included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
months | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. | NA [8.80 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure.

6. Primary Outcome: Overall Survival (OS)
Description: OS was defined as time from first dose of belumosudil to the date of death due to any cause. CI was calculated using Kaplan-Meier method.
Time Frame: From first dose of study drug (Day 1) to the date of death due to any cause, up to approximately 24 months
Population: The full analysis set included all participants enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Belumosudil 400 mg QD: Participants received belumsudil 400 mg tablet orally QD until cGVHD progression, unacceptable toxicity or up to 2 years at the discretion of the Investigator.
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
months | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure. | NA [NA to NA] — NA indicates that median, lower and upper limit of CI were not estimable due to insufficient number of participants with events at study closure.

7. Primary Outcome: Percentage of Participants With Complete Response (CR) and Partial Response (PR)
Description: As per the 2014 NIH Consensus Development Project for clinical trials in cGVHD criteria: CR was defined as resolution of all manifestations of cGVHD in each organ or site. PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: At Baseline (Day 1), Month 3 and every 3 months thereafter (+/-14 days), up to 23 months
Population: The full analysis set included all participants enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
percentage of participants
  CR | 30.8 | 11.1 | 0
  PR | 30.8 | 77.8 | 0

8. Primary Outcome: Number of Participants With Best Response by Organ System
Description: The best response (CR, PR) for individual organs (skin, eyes, mouth, esophagus, upper gastrointestinal [GI], lower GI, liver, lungs, joints and fascia) was summarized. As per the 2014 NIH Consensus Development Project for clinical trials in cGVHD criteria, CR was defined as resolution of all manifestations of cGVHD in each organ or site. PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site.
Time Frame: At Baseline (Day 1), Month 3 and every 3 months thereafter (+/-14 days), up to 23 months
Population: The full analysis set included all participants enrolled in the study. Only those participants with data collected for each specified category are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 10 | 8 | 1
Participants
  Skin: number analyzed (Participants) | 9 | 8 | 1
  Skin | 6 | 5 | 0
  Eyes | 6 | 4 | 0
  Mouth: number analyzed (Participants) | 6 | 4 | 1
  Mouth | 4 | 3 | 0
  Esophagus: number analyzed (Participants) | 1 | 3 | 0
  Esophagus | 1 | 2 | 0
  Upper GI: number analyzed (Participants) | 0 | 1 | 0
  Upper GI | 0 | 0 | 0
  Lower GI: number analyzed (Participants) | 1 | 1 | 0
  Lower GI | 0 | 1 | 0
  Liver: number analyzed (Participants) | 2 | 0 | 0
  Liver | 1 | 0 | 0
  Lungs: number analyzed (Participants) | 5 | 3 | 1
  Lungs | 1 | 3 | 0
  Joints and Fascia: number analyzed (Participants) | 8 | 8 | 0
  Joints and Fascia | 5 | 7 | 0

9. Primary Outcome: Percent Change From Baseline in Corticosteroid Dose to Greatest Reduction
Description: Change in corticosteroid doses was analyzed by using prednisone dose equivalents. If participants were not using prednisone as the systemic corticosteroid, then the prednisone dose equivalent would be determined according to following conversion ratios: 1 mg prednisone is equivalent to: 4.0 mg Hydrocortisone; 0.8 mg Methylprednisolone; 0.15 mg Dexamethasone; 1.0 mg Prednisolone and 0.8 mg Triamcinolone. Baseline was defined as the valid and last non-missing value obtained within 28 days prior to participant receiving the first study drug in parent study (KD025-208 [NCT02841995] or KD025-213 [NCT03640481]).
Time Frame: Baseline (Day 1) and Month 23
Population: The full analysis set included all participants enrolled in the study. Only those participants with data collected at specified timepoints are reported.
Measure: Median (Full Range); unit: percent change
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 4 | 2 | 0
percent change | -50.00 [-100.00 to 0.0] | 0.0 [0.0 to 0.0] |

10. Primary Outcome: Number of Participants With Maximal Improvement From Baseline in Global Severity Rating (GSR) Based on Clinician-Reported Chronic Graft-Versus-Host-Disease Assessment
Description: The GSR assessment was performed by asking the participants to rate their disease severity of cGVHD symptoms on a 0 to 10-point numeric rating scale, where score 0 indicated 'not at all severe cGVHD symptoms' and score 10 indicated 'most severe cGVHD symptoms possible'. The response was defined using scores from 9 organs: skin, eyes, mouth, esophagus, upper GI track, lower GI tract, liver, lungs, and joints and fascia plus GSR. Baseline was defined as the valid and last non-missing value obtained within 28 days prior to participant receiving the first study drug in parent study (KD025-208 [NCT02841995] or KD025-213 [NCT03640481]). Maximal improvement from Baseline was calculated as lowest GSR score on scheduled visits minus GSR score at Baseline with possible ranges from -10 to 10. The lower the number means the better improvement in cGVHD symptoms.
Time Frame: From Baseline (Day 1) up to 23 months
Population: The full analysis set included all participants enrolled in the study. Only those categories in which at least 1 participant had data are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
Participants
  -8 | 1 | 1 | 0
  -7 | 0 | 1 | 0
  -6 | 3 | 0 | 0
  -5 | 2 | 2 | 0
  -4 | 0 | 1 | 0
  -3 | 1 | 1 | 0
  -2 | 1 | 1 | 0
  -1 | 1 | 1 | 0
  0 | 1 | 0 | 0

11. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), Grade >=3 Treatment-Emergent Adverse Events and Deaths
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant associated with the use of a study drug, whether or not considered drug-related. Serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, was a congenital anomaly/birth defect or was an important medical event. The severity of each AE was graded using the Common Terminology Criteria for Adverse Events version 4.03 scale. TEAEs were defined as AEs that developed, worsened or became serious during the TE period.
Time Frame: From the first dose of study drug (Day 1) up to 28 days after the last dose of study drug, approximately 24 months
Population: The full analysis set included all participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
Number analyzed (Participants) | 13 | 9 | 1
Participants
  TEAEs | 8 | 7 | 0
  TESAEs | 4 | 2 | 0
  Grade >=3 TEAEs | 3 | 4 | 0
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (Day 1) up to 28 days after the last dose of study drug, approximately 24 months
Description: Analysis was performed on the full analysis set.
Arm/Group | Belumosudil 200 mg QD | Belumosudil 200 mg BID | Belumosudil 400 mg QD
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/1
Serious Adverse Events (participants affected / at risk) | 4/13 | 2/9 | 0/1
Other Adverse Events (participants affected / at risk) | 8/13 | 7/9 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil 200 mg QD (N=13) | Belumosudil 200 mg BID (N=9) | Belumosudil 400 mg QD (N=1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dacryoadenitis Acquired (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue Dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil 200 mg QD (N=13) | Belumosudil 200 mg BID (N=9) | Belumosudil 400 mg QD (N=1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemophilus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis Externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Intraductal Papillary-Mucinous Carcinoma Of Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior Vena Cava Syndrome (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Nasal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oral Dysaesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nonalcoholic Fatty Liver Disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Tightness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Hydrometra (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood Glucose Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT05305989/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT05305989/SAP_001.pdf